CLINICAL TRIAL: NCT01309373
Title: Epidemiological Study to Assess the Psychosocial and Symptomatic Remission and Community Integration Status in Patients With Schizophrenia (REINTEGRA Study)
Brief Title: An Epidemiological Study to Assess the Psychosocial and Symptomatic Remission and Community Integration Status in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR016684; RISSCH4248 (Other: Janssen-Cilag S.A., Spain)
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; Schizoaffective Disorder; Remission; Psychosocial; Symtomatic; Integration; Schizoaffective; Adherence
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Patient Outcome Assessment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Patient assessment 2 scales will be used to assesss the remission of schizophrenia (APA scale and PSRS scale). The BPRS scale will be used to assess the clinical integration of patients.
  Interventions: Other: Patient assessment

INTERVENTIONS:
Other: Patient assessment — 2 scales will be used to assesss the remission of schizophrenia (APA scale and PSRS scale). The BPRS scale will be used to assess the clinical integration of patients.

SUMMARY:
The purpose of this study is to estimate the level of symptomatic and psychosocial remission of patients with schizophrenia and schizoaffective disorder in standard clinical practice as a function of the degree of adherence to antipsychotic treatment. The secondary objectives are to study the level of community integration of the patients included in the study, and its influencing factors, to analyze the role of various sociodemographic factors, factors related to the course of disease and the psychopathological status of the patient in community integration and remission, to analyze the potential predictors of a favorable course (symptomatic and psychosocial remission) and a poor course (no symptomatic or psychosocial remission), to assess the impact of treatment adherence on the change in the functional and community integration status of patients (based on the occupation, independence level, and degree of disability variables), to assess the significance of premorbid (academic and social) adjustment in the symptomatic and functional remission and the community integration status of patients and to correlate the level of insight to the remission and integration status of patients.

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional, non-interventional observational, cohort epidemiological study conducted in the outpatient mental health facility setting in patients with schizophrenia. The inclusion of two patient cohorts is contemplated, recruited in mental health facilities. One cohort will involve patients estimated to have inadequate adherence to antipsychotic treatment, while the other will consist of patients with adequate adherence to such treatment. N/A

ELIGIBILITY:
Inclusion Criteria:

* Patients with schizophrenia or schizoaffective disorder being followed-up at a mental health facility
* Whose clinical records of recent years may be accessed
* Who has signed informed consent, stating that he/she understands the study purpose and requirements and gives consent to participate in the study
* In whom the psychiatrist and main caregiver may estimate the degree of adherence to antipsychotic treatment during the last two years
* Not hospitalized in acute disorder units in the last 12 months

Exclusion Criteria:

* Patients with psychiatric disease other than schizophrenia or schizoaffective disorder who have been diagnosed with severe to moderate mental retardation, organic disorders of personality, and/or severe and/or disabling neurological disease
* Patients who are actively participating in any clinical trial/study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in Spanish outpatient mental health facilities, with schizophrenia or schizoaffective disorder
Sampling Method: Probability Sample
Enrollment: 1809 (Actual)
Dates: Start 2010-11; Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.